CLINICAL TRIAL: NCT06143592
Title: The Effect of Inspiratory Muscle Training on Balance, Falls and Diaphragm Thickness in the Elderly: A Randomized Controlled Trial
Brief Title: Inspiratory Muscle Training on Balance, Falls and Diaphragm Thickness in the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ekin TACALAN, MSc, PT, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Inspiratory Muscle Training
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Sarcopenia
Keywords: falls; exercise; elderly
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-Intensity Inspiratory Muscle Training Group (LI-IMT) (Experimental): Before the training, the MIP value is recorded in "cmH2O". The inspiratory muscle training intensity in the first four weeks is determined by taking 30% of the MIP value and the resistance of the device is adjusted to this level. The pressure measurements of the participants are repeated in the 4th week and the new MIP value is determined. Then, 30% of the new MIP value is taken to determine the training intensity in the 4th to 8th week and the resistance of the device is adjusted to this new level. This situation is repeated in the same way in the 8th week and the new training intensity in the 8th to 12th week is determined by taking 30% of the new MIP value. According to the MIP values obtained during the entire training period, participants are asked to work at home for 12 weeks, three to five days a week, 2 times a day, 15-minutes each, 30 minutes total.
  Interventions: Other: Inspiratory Muscle Training
- Modarate-Intensity Inspiratory Muscle Training Group (MI-IMT) (Experimental): Before the training, the MIP value is recorded in "cmH2O". The inspiratory muscle training intensity in the first four weeks is determined by taking 50% of the MIP value and the resistance of the device is adjusted to this level. The pressure measurements of the participants are repeated in the 4th week and the new MIP value is determined. Then, 50% of the new MIP value is taken to determine the training intensity in the 4th to 8th week and the resistance of the device is adjusted to this new level. This situation is repeated in the same way in the 8th week and the new training intensity in the 8th to 12th week is determined by taking 50% of the new MIP value. According to the MIP values obtained during the entire training period, participants are asked to work at home for 12 weeks, three to five days a week, 2 times a day, 15-minutes each, 30 minutes total.
  Interventions: Other: Inspiratory Muscle Training
- Control Group (Sham Group) (Experimental): Participants in the control group are given a POWERbreathe® device with the resistance set to the lowest level (0 cmH2O) at the end of the session where the initial assessments are made. As in the training group, participants are asked to work at home for 12 weeks, three to five days a week, 2 times a day, 15-minutes each, 30 minutes total. In order to eliminate the learning effect on the participants, pressure measurements are made in the 4th and 8th weeks, but the training intensity is kept constant at the lowest level during the 12 weeks.
  Interventions: Other: Inspiratory Muscle Training

INTERVENTIONS:
Other: Inspiratory Muscle Training — Inspiratory muscle training is performed using POWERbreathe® (Powerbreathe, POWERbreathe International Ltd.Warwickshire, England) with a working range of 10-90 cmH2O with the inspiratory threshold pressure loading method. The device is given to each participant to use at home, so Gazi University Scientific Research Projects Coordination Unit (BAP) was applied for the supply of the devices. At the end of the session in which the initial evaluations of all participants are made, the participants are told how to work with the device, the resistance levels of the device and the points to be considered during the application. A sample application session is performed with the participants under the supervision of a specialist physiotherapist. Participants are called by the same physiotherapist every two days by phone to ensure their compliance with the training.

SUMMARY:
Decreases in body muscle mass, function and strength occur with ageing and this condition is called "sarcopenia". It is known that sarcopenic elderly people fall more than non-sarcopenic elderly people, their balance is negatively affected, their diaphragm thickness decreases and their quality of life may decrease due to their lower functional capacity. Although exercise training, which is considered among the approaches in the treatment of sarcopenia, has been shown to be an effective method, the effects of inspiratory muscle training applied at different intensities are relatively limited. Therefore, in this study, we are investigating the effects of low [30% of maximal inspiratory pressure (MIP)] and moderate (50% of MIP) inspiratory muscle training on respiratory and peripheral muscle strength, physical performance, functional capacity, balance, fear of falling, quality of life, diaphragm thickness and stiffness in sarcopenic elderly. In this study, participants are randomly divided into 3 groups: a low-intensity inspiratory muscle training group, a moderate-intensity inspiratory muscle training group and control (sham) group by simple random method after being evaluated for respiratory and peripheral muscle strength, physical performance, functional capacity, balance, fear of falling, quality of life, diaphragm thickness and stiffness.

DETAILED DESCRIPTION:
INTRODUCTION

The proportion of the elderly population compared to the total population is increasing worldwide. While this rate was 8.3% in 2015, it is predicted to reach 17.8% by 2060. Decreases in body muscle mass, function and strength occur with ageing and this condition is called "sarcopenia". The European Working Group on Sarcopenia in Older People (EWGSOP) defined sarcopenia as a syndrome characterized by a loss not only in muscle mass but also in muscle strength or physical performance, leading to movement disorders, hospitalization and falls. In studies, it was found that the frequency of falls in sarcopenic participants was higher than in non-sarcopenic participants. In addition, it has been shown that sarcopenia negatively affects balance in the elderly, sarcopenic participants have shorter standing times on one leg compared to non-sarcopenic participants, their diaphragm thickness decreases and their quality of life decreases due to their lower functional capacity.

In order to make a diagnosis of sarcopenia, the current situation of the participant should be analyzed in terms of "muscle mass", "muscle strength" and "physical performance". Methods such as Magnetic Resonance, Dual Energy X-ray Absorptiometry (DEXA), Computed Tomography, Bioimpedance Analysis (BIA), and circumference measurement are preferred in the evaluation of muscle mass; dynamometer is preferred in the evaluation of muscle strength; and tests such as walking speed, timed get up and go test, sit up and stand test from a chair are preferred in the evaluation of physical performance. Important approaches in the prevention and treatment of sarcopenia are exercise, physical activity and nutritional support. Exercise training in the treatment of sarcopenia has been shown to be an effective method to increase muscle mass and strength in the elderly. Both aerobic and resistance exercises have been shown to decrease the rate of decline in muscle mass and increase endurance with age. The literature shows that studies have focused especially on exercises involving peripheral muscles. However, sarcopenia may affect respiratory muscles in addition to peripheral muscles.

Respiratory muscle training is a specific exercise training applied to respiratory muscles using skeletal muscle training principles in order to increase respiratory muscle strength and endurance, correct the length-tension relationship of respiratory muscles and increase respiratory capacity. The most common approach to respiratory muscle training is the inspiratory threshold pressure loading method. In the only study in the literature to our knowledge that examined the effect of inspiratory muscle training in sarcopenic elderly, the authors compared the effect of peripheral and respiratory exercises on isometric knee extension and arm flexion strength, hand grip strength, inspiratory and expiratory muscle strength and walking speed, but did not examine the effect of training on functional capacity, balance, fear of falling, quality of life, diaphragm thickness and stiffness.

Studies on inspiratory muscle training in elderly participants have shown an increase in functional capacity and exercise capacity, improvement in inspiratory muscle strength and expiratory muscle strength, improvement in balance and physical performance, increase in diaphragm thickness, improvement in lower extremity muscle strength and improvement in quality of life; however, in the systematic review published in 2020 on inspiratory muscle training in the elderly, it was emphasized that the intensity of training (maximal inspiratory pressure-MIP) varies between 30% and 80%, and there is no consensus in the literature on loading. The effect of inspiratory muscle training at different intensities in a healthy elderly population was investigated for the first time by Martin-Sanchez et al. (2020), who emphasized the effectiveness of exercise performed at 20% and 40% of MIP. However, since there is no study to our knowledge on inspiratory muscle training applied at different intensities in sarcopenic elderly, our study will investigate the effects of low (30% of MIP) and moderate (50% of MIP) intensity inspiratory muscle training on respiratory and peripheral muscle strength, physical performance, functional capacity, balance, fear of falling, quality of life, diaphragm thickness and stiffness in sarcopenic elderly.

METHODS

Design:

Participants aged 65 years and over diagnosed with sarcopenia by the relevant physician in Gazi University Faculty of Medicine, Department of Internal Medicine, Geriatrics Division Outpatient Clinic are included. In this randomized controlled single-blind study, the participants are randomly divided into 3 groups: low-intensity inspiratory muscle training group, moderate-intensity inspiratory muscle training group and control (sham) group by simple random method after being evaluated. The evaluations are performed face to face at Gazi University Faculty of Medicine, Department of Internal Medicine, Division of Geriatrics. Except for respiratory muscle strength assessment, participants in the treatment group will be evaluated at baseline and at the 12th week after treatment; participants in the control group will be evaluated at baseline and at the end of the 12th week; respiratory muscle strength will be evaluated at baseline, at week 4, at week 8 and at week 12 in all groups. The Ethics Committee of Gazi University provided ethical approval (2022-19/12.12.2022). All participants included in the study will read and sign the written informed consent form prior to evaluation according to the principles of the Declaration of Helsinki. The rights of the participants are fully protected during the study procedures.

Sample Size:

In line with a similar study in the literature, using G*power software (version 3.1, Universitat Düsseldorf, Germany), the number of participants required to reach a power level of 0.80 at 5% type 1 error level with an effect size of 0.60 was determined as 30 participants.

Randomization and Blinding:

Before enrolment in the study, patients are randomly assigned to 3 groups according to an online randomization table (https://www.random.org, 2023-03-27, 11:16:08 UTC). The randomization program is computer-generated using a basic random number generator in blocks. Participants are blinded to the intervention groups that they are assigned to.

Statistical Analysis:

IBM SPSS Statistics 25 (Statistical Package for the Social Sciences) analysis program will be used for statistical analysis. Descriptive analyses will be calculated with minimum-maximum, mean±standard deviation (X±SD) and median (interquartile range-IQR) for numerical data. For categorical data, number (n) and percentage (%) values will be defined. The suitability of the data obtained from participants to normal distribution will be evaluated by Skewness, Kurtosis, Histogram Analysis, Kolmogorov-Smirnov Test and coefficient of variation ratio. The difference between the change in measurement values of participants according to the intervention programs will be calculated by ANOVA one-way analysis of variance if the data fits the normal distribution, and by Kruskal Wallis-H Test if the data does not fit the normal distribution. Post-hoc tests will be applied to investigate the differences between the groups.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with sarcopenia,
* 65 years of age or older,
* scoring above 21 on the Mini-Mental State Scale,
* volunteering to participate in the study.

Exclusion Criteria:

* active smoker or quit smoking in less than 5 years,
* undergone abdominal surgery, thoracic surgery or lower extremity surgery,
* fracture within the last 1 year,
* having a condition that prevents bioelectrical impedance measurement such as pacemaker, implant,
* having a disease such as pulmonary artery hypertension, glaucoma, an aneurysm that prevents the Valsalva manoeuvre,
* having hypertension that cannot be controlled with antihypertensive medication,
* having a neurological disease affecting mobility such as cerebrovascular disease, Parkinson's disease,
* having chronic inflammatory disease known to affect muscle metabolism, including uncontrolled diabetes (Hba1c>9), rheumatoid arthritis,
* presence of any acute and chronic cardiovascular disease such as unstable angina pectoris, recent myocardial infarction, uncontrolled cardiac arrhythmia, congestive heart failure, acute ischemic heart disease,
* presence of any acute and chronic pulmonary disease such as COPD, acute pulmonary embolism, pulmonary oedema,
* having a history of cancer.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Respiratory Muscle Strength Assessment | at baseline, at week 4, at week 8, at week 12
  The easiest and most commonly used method to measure respiratory muscle strength is maximal inspiratory and expiratory pressure measurements. Maximal inspiratory pressure (MIP) indicates inspiratory muscle strength. Maximal expiratory pressure (MEP) reflects expiratory muscle strength. Standard guidelines set by the American Thoracic Society/European Respiratory Society will be followed during the assessments. For the MIP assessment, the participant will be asked to perform a maximal expiration manoeuvre followed by maximal inspiration for 1-3 seconds (Müller manoeuvre). For the MEP assessment, the participant first performs a maximum inspiration manoeuvre, followed by maximum expiration for 1-3 seconds (Valsalva manoeuvre). In our study, measurements will be performed with a mobile and easy-to-use electronic pressure measuring device (MicroRPM, Vyaire Medical, Mettawa, IL).
Peripheral Muscle Strength Assessment: Hand Grip Strength | at baseline and at the end of 12th week
  Hand grip strength is a reliable method that provides information about upper extremity muscle strength in elderly participants. A hand dynamometer (Jamar, Fabrication Enterprised Inc., Irvington, New York) will be used in the evaluation. The measurements are made in the test position standardized by the American Association of Hand Therapists with the tested arm sitting upright in an unsupported chair with the shoulder in adduction, elbow in 90º flexion, forearm in neutral position, wrist in 0-30º extension and 0-15º ulnar deviation. During the assessment, the participant is asked to squeeze the dynamometer with all his/her strength and then let his/her hand go completely relaxed. This process is performed three times and the average of these values is recorded in kg/force. In our study, hand grip strength will be measured for both hands.
Peripheral Muscle Strength Assessment: Knee Extension Strength | at baseline and at the end of 12th week
  Knee extension strength will be measured with a manual muscle tester (Lafayette Instrument Company, Lafayette, Indiana) in a sitting position with the hip and knee joint in 90° flexion. During the measurement from the distal tibia, the participant is asked to bring the knee to full extension. Each measurement is performed three times and muscle strength is determined by taking the arithmetic mean of the total value. In our study, knee extension strength will be measured for both legs.
Dynamic Balance Assessment: Mini-Balance Evaluation Systems Test (Mini-BESTest) | at baseline and at the end of 12th week
  Participants' dynamic balance will be assessed using the Mini BESTest, the short version of BESTest. The questionnaire, which consists of 14 items in total, has 4 sub-items in total, including anticipatory postural control (standing up from a sitting position, standing on tiptoe, standing on one leg), reactive postural control (forward, backward and lateral compensatory corrective stepping), sensory orientation (firm surface with eyes open, foam surface with eyes closed and inclined surface with eyes closed), dynamic gait (change in gait speed, walking with horizontal head movements, pivoting while walking, stepping over obstacles, timed stand and walk with double task). The score of each item ranges from "0" to "2" and the total score ranges from "0" to "28". A high score indicates good balance.
Diaphragm Thickness and Stiffness Assessment | at baseline and at the end of 12th week
  Diaphragm thickness and stiffness will be evaluated by the relevant physician using an ultrasound device. The probe will be placed between the anterior and middle axillary lines of the 9th or 10th intercostal spaces while the participant is in the supine position. Assessments will be performed during the peak inspiration and end-expiration phases of the normal respiratory cycle.
Static Balance Asssesment | at baseline and at the end of 12th week
  Static balance measurements of participants will be performed with Biodex Balance System® (Biodex Medical Systems, Inc., United States of America). With this balance device, "postural stability", "limits of stability" and "fall risk" of participants are evaluated. All tests will be performed bipedal with bare feet on a standard support surface.
Static Balance Asssesment: Postural Stability Test | at baseline and at the end of 12th week
  In this test, participants will be instructed to stand still on the platform and the displacement of the centre of gravity (COG) is quantified for anterior-posterior (AP) and medial-lateral (ML) axes. It gives three types of outcome measures: overall stability index, AP stability index and ML stability index. Higher scores indicate worse postural stability. In our study, the test will be repeated three times for 30 seconds and 10 seconds rest will be given between repetitions.
Static Balance Asssesment: Limits of Stability Test | at baseline and at the end of 12th week
  This test tests the participant's ability to control and move the centre of gravity within the limits of the support surface. The difficulty level of the test is "easy", "medium", "difficult". The participant is asked to reach out in a linear fashion by shifting the centre of gravity towards the ball in eight different directions flashing on the screen. This is repeated three times with a 10-second rest between repetitions. Low scores express poor postural control. In our study, the "easy" test will be applied, and the completion time of the test, the percentage score of stability in each direction and the total percentage score will be used in the data analysis of our study.
Static Balance Asssesment: Modified Balance Sensory Integration Test | at baseline and at the end of 12th week
  In our study, this test will be used to assess the fall risk of participants. The participant is asked to stand upright with both feet shoulder-width apart and hands at the sides, in the most comfortable position to maintain balance. The test is administered in four different situations: firm surface with eyes open/closed, foam surface with eyes open/closed. The device gives the sway index score of the participant in these four different situations. A higher sway index score indicates increased postural sway. In our study, the test will be repeated three times for 30 seconds and 10 seconds rest will be given between repetitions.

SECONDARY OUTCOMES:
Physical Performance Assessment: Timed Get Up and Go Test | at baseline and at the end of 12th week
  Developed in 1991 by Podsiadlo and Richardson, this test aims to assess balance and mobility and is an objective, reliable and simple test. The participant is expected to get up from the chair, walk 3 meters, turn around, return to the chair and sit on the chair again. The time it takes the participant to complete the test is recorded.
Physical Performance Assessment: Sit up and Stand Test from a Chair | at baseline and at the end of 12th week
  The test starts in a sitting position. The participant sits on a chair with hands crossed over the chest. Duration in seconds is held. The participant gets up and down from the chair five times as fast as possible. The test is terminated on the last rise. The test is performed twice. The best score is recorded.
Functional Capacity Assessment: Six Minute Walk Test | at baseline and at the end of 12th week
  Developed in 1963 by Balke to measure functional capacity, this test measures the distance in meters a participant can walk in six minutes on a flat surface, as fast as possible but without running. The participant is told that if he/she feels respiratory problems such as shortness of breath during the application, he/she can decrease his/her speed and rest, but the elapsed time will be included in the test. A 30-meter-long walking area is determined for the test, turning points are marked and care is taken to ensure no obstacles and crowds are on the track. At the end of the test, measurements are repeated and the distance walked is recorded in meters.
Fear of Falling Assessment: Falls Efficacy Scale International (FES-I) | at baseline and at the end of 12th week
  This scale, developed by Yardley et al. (2005) to assess the fear of falling in participants, assesses how confident older people are in their activities of daily living and indicates the level of fall concerns. The scale consists of 16 items, each rated on a 4-point scale. The total score range is from 16 (no worry about falling) to 64 (extreme worry about falling). A score between 16-19 indicates a "low fear of falling", a score between 20-27 indicates a "moderate fear of falling" and a score between 28-64 indicates a "high fear of falling". The Turkish validity and reliability of the scale was conducted by Ulus et al. (2012).
Quality of Life Assessment: Sarcopenia Quality of Life Questionnaire (SarQoL) | at baseline and at the end of 12th week
  This questionnaire developed by Beaudart et al. (2015) consists of 22 questions with 55 items. It consists of 7 sub-parameters including "physical and mental health, movement, body composition, functionality, activities of daily living, leisure time activities and fears". The total score ranges from 0 (worst health) to 100 (best health). The Turkish validity and reliability study of the questionnaire was conducted by Erdoğan et al. (2021).

CONTACTS AND LOCATIONS:
Overall Officials: Selda Başar, Study Director — Gazi University
Locations (1):
- Ankara Dr. Sami Ulus Children Health and Diseases Training and Research Hospital, Ankara, Altındağ/Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kato K, Hatanaka Y. The influence of trunk muscle strength on walking velocity in elderly people with sarcopenia. J Phys Ther Sci. 2020 Feb;32(2):166-172. doi: 10.1589/jpts.32.166. Epub 2020 Feb 14. PMID 32158081
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Aibar-Almazan A, Martinez-Amat A, Cruz-Diaz D, Jimenez-Garcia JD, Achalandabaso A, Sanchez-Montesinos I, de la Torre-Cruz M, Hita-Contreras F. Sarcopenia and sarcopenic obesity in Spanish community-dwelling middle-aged and older women: Association with balance confidence, fear of falling and fall risk. Maturitas. 2018 Jan;107:26-32. doi: 10.1016/j.maturitas.2017.10.001. Epub 2017 Oct 7. PMID 29169576
- [Background] Gadelha AB, Neri SGR, Oliveira RJ, Bottaro M, David AC, Vainshelboim B, Lima RM. Severity of sarcopenia is associated with postural balance and risk of falls in community-dwelling older women. Exp Aging Res. 2018 May-Jun;44(3):258-269. doi: 10.1080/0361073X.2018.1449591. Epub 2018 Mar 20. PMID 29558320
- [Background] Bouchard DR, Dionne IJ, Brochu M. Sarcopenic/obesity and physical capacity in older men and women: data from the Nutrition as a Determinant of Successful Aging (NuAge)-the Quebec longitudinal Study. Obesity (Silver Spring). 2009 Nov;17(11):2082-8. doi: 10.1038/oby.2009.109. Epub 2009 Apr 16. PMID 19373219
- [Background] Deniz O, Coteli S, Karatoprak NB, Pence MC, Varan HD, Kizilarslanoglu MC, Oktar SO, Goker B. Diaphragmatic muscle thickness in older people with and without sarcopenia. Aging Clin Exp Res. 2021 Mar;33(3):573-580. doi: 10.1007/s40520-020-01565-5. Epub 2020 May 13. PMID 32406014
- [Background] Yuenyongchaiwat K, Akekawatchai C. Systemic Inflammation in Sarcopenia Alter Functional Capacity in Thai Community-dwelling Older People: A Preliminary Observational Study. Curr Aging Sci. 2022 Aug 4;15(3):274-281. doi: 10.2174/1874609815666220513141300. PMID 35570546
- [Background] Yu S, Umapathysivam K, Visvanathan R. Sarcopenia in older people. Int J Evid Based Healthc. 2014 Dec;12(4):227-43. doi: 10.1097/XEB.0000000000000018. PMID 25478672
- [Background] Giallauria F, Cittadini A, Smart NA, Vigorito C. Resistance training and sarcopenia. Monaldi Arch Chest Dis. 2016 Jun 22;84(1-2):738. doi: 10.4081/monaldi.2015.738. PMID 27374049
- [Background] Frankel JE, Bean JF, Frontera WR. Exercise in the elderly: research and clinical practice. Clin Geriatr Med. 2006 May;22(2):239-56; vii. doi: 10.1016/j.cger.2005.12.002. PMID 16627076
- [Background] Martin Del Campo Cervantes J, Habacuc Macias Cervantes M, Monroy Torres R. Effect of a Resistance Training Program on Sarcopenia and Functionality of the Older Adults Living in a Nursing Home. J Nutr Health Aging. 2019;23(9):829-836. doi: 10.1007/s12603-019-1261-3. PMID 31641732
- [Background] Cebria I Iranzo MA, Balasch-Bernat M, Tortosa-Chulia MA, Balasch-Parisi S. Effects of Resistance Training of Peripheral Muscles Versus Respiratory Muscles in Older Adults With Sarcopenia Who are Institutionalized: A Randomized Controlled Trial. J Aging Phys Act. 2018 Oct 1;26(4):637-646. doi: 10.1123/japa.2017-0268. Epub 2018 Aug 27. PMID 29431561
- [Background] Lotters F, van Tol B, Kwakkel G, Gosselink R. Effects of controlled inspiratory muscle training in patients with COPD: a meta-analysis. Eur Respir J. 2002 Sep;20(3):570-6. doi: 10.1183/09031936.02.00237402. PMID 12358330
- [Background] Gosselink R, De Vos J, van den Heuvel SP, Segers J, Decramer M, Kwakkel G. Impact of inspiratory muscle training in patients with COPD: what is the evidence? Eur Respir J. 2011 Feb;37(2):416-25. doi: 10.1183/09031936.00031810. PMID 21282809
- [Background] Aznar-Lain S, Webster AL, Canete S, San Juan AF, Lopez Mojares LM, Perez M, Lucia A, Chicharro JL. Effects of inspiratory muscle training on exercise capacity and spontaneous physical activity in elderly subjects: a randomized controlled pilot trial. Int J Sports Med. 2007 Dec;28(12):1025-9. doi: 10.1055/s-2007-965077. Epub 2007 May 29. PMID 17534784
- [Background] Rodrigues GD, Gurgel JL, Goncalves TR, da Silva Soares PP. Inspiratory muscle training improves physical performance and cardiac autonomic modulation in older women. Eur J Appl Physiol. 2018 Jun;118(6):1143-1152. doi: 10.1007/s00421-018-3844-9. Epub 2018 Mar 16. PMID 29549494
- [Background] Ferraro FV, Gavin JP, Wainwright T, McConnell A. The effects of 8 weeks of inspiratory muscle training on the balance of healthy older adults: a randomized, double-blind, placebo-controlled study. Physiol Rep. 2019 May;7(9):e14076. doi: 10.14814/phy2.14076. PMID 31074198
- [Background] Mills DE, Johnson MA, Barnett YA, Smith WH, Sharpe GR. The effects of inspiratory muscle training in older adults. Med Sci Sports Exerc. 2015 Apr;47(4):691-7. doi: 10.1249/MSS.0000000000000474. PMID 25116085
- [Background] Martin-Sanchez C, Barbero-Iglesias FJ, Amor-Esteban V, Martin-Nogueras AM. Comparison between Two Inspiratory Muscle Training Protocols, Low Loads versus High Loads, in Institutionalized Elderly Women: A Double-Blind Randomized Controlled Trial. Gerontology. 2021;67(1):1-8. doi: 10.1159/000511009. Epub 2020 Dec 17. PMID 33333521
- [Background] Souza H, Rocha T, Pessoa M, Rattes C, Brandao D, Fregonezi G, Campos S, Aliverti A, Dornelas A. Effects of inspiratory muscle training in elderly women on respiratory muscle strength, diaphragm thickness and mobility. J Gerontol A Biol Sci Med Sci. 2014 Dec;69(12):1545-53. doi: 10.1093/gerona/glu182. PMID 25395284
- [Background] Seixas MB, Almeida LB, Trevizan PF, Martinez DG, Laterza MC, Vanderlei LCM, Silva LP. Effects of Inspiratory Muscle Training in Older Adults. Respir Care. 2020 Apr;65(4):535-544. doi: 10.4187/respcare.06945. Epub 2019 Oct 29. PMID 31662444
- [Background] Black LF, Hyatt RE. Maximal respiratory pressures: normal values and relationship to age and sex. Am Rev Respir Dis. 1969 May;99(5):696-702. doi: 10.1164/arrd.1969.99.5.696. No abstract available. PMID 5772056
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Dodds RM, Syddall HE, Cooper R, Benzeval M, Deary IJ, Dennison EM, Der G, Gale CR, Inskip HM, Jagger C, Kirkwood TB, Lawlor DA, Robinson SM, Starr JM, Steptoe A, Tilling K, Kuh D, Cooper C, Sayer AA. Grip strength across the life course: normative data from twelve British studies. PLoS One. 2014 Dec 4;9(12):e113637. doi: 10.1371/journal.pone.0113637. eCollection 2014. PMID 25474696
- [Background] Sipers WM, Verdijk LB, Sipers SJ, Schols JM, van Loon LJ. The Martin Vigorimeter Represents a Reliable and More Practical Tool Than the Jamar Dynamometer to Assess Handgrip Strength in the Geriatric Patient. J Am Med Dir Assoc. 2016 May 1;17(5):466.e1-7. doi: 10.1016/j.jamda.2016.02.026. PMID 27107163
- [Background] Francis P, Toomey C, Mc Cormack W, Lyons M, Jakeman P. Measurement of maximal isometric torque and muscle quality of the knee extensors and flexors in healthy 50- to 70-year-old women. Clin Physiol Funct Imaging. 2017 Jul;37(4):448-455. doi: 10.1111/cpf.12332. Epub 2016 Jan 7. PMID 26749301
- [Background] Arnold BL, Schmitz RJ. Examination of balance measures produced by the biodex stability system. J Athl Train. 1998 Oct;33(4):323-7. PMID 16558529
- [Background] Clark S, Rose DJ, Fujimoto K. Generalizability of the limits of stability test in the evaluation of dynamic balance among older adults. Arch Phys Med Rehabil. 1997 Oct;78(10):1078-84. doi: 10.1016/s0003-9993(97)90131-3. PMID 9339156
- [Background] Cohen H, Blatchly CA, Gombash LL. A study of the clinical test of sensory interaction and balance. Phys Ther. 1993 Jun;73(6):346-51; discussion 351-4. doi: 10.1093/ptj/73.6.346. PMID 8497509
- [Background] Franchignoni F, Horak F, Godi M, Nardone A, Giordano A. Using psychometric techniques to improve the Balance Evaluation Systems Test: the mini-BESTest. J Rehabil Med. 2010 Apr;42(4):323-31. doi: 10.2340/16501977-0537. PMID 20461334
- [Background] Sendur HN, Cerit MN, Sendur AB, Ozhan Oktar S, Yucel C. Evaluation of Diaphragm Thickness and Stiffness Using Ultrasound and Shear-Wave Elastography. Ultrasound Q. 2022 Jan 10;38(1):89-93. doi: 10.1097/RUQ.0000000000000593. PMID 35001026
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Yelnik A, Bonan I. Clinical tools for assessing balance disorders. Neurophysiol Clin. 2008 Dec;38(6):439-45. doi: 10.1016/j.neucli.2008.09.008. Epub 2008 Oct 18. PMID 19026963
- [Background] BALKE B. A SIMPLE FIELD TEST FOR THE ASSESSMENT OF PHYSICAL FITNESS. REP 63-6. Rep Civ Aeromed Res Inst US. 1963 Apr:1-8. No abstract available. PMID 14131272
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Burr JF, Bredin SS, Faktor MD, Warburton DE. The 6-minute walk test as a predictor of objectively measured aerobic fitness in healthy working-aged adults. Phys Sportsmed. 2011 May;39(2):133-9. doi: 10.3810/psm.2011.05.1904. PMID 21673494
- [Background] Yardley L, Beyer N, Hauer K, Kempen G, Piot-Ziegler C, Todd C. Development and initial validation of the Falls Efficacy Scale-International (FES-I). Age Ageing. 2005 Nov;34(6):614-9. doi: 10.1093/ageing/afi196. PMID 16267188
- [Background] Ulus Y, Durmus D, Akyol Y, Terzi Y, Bilgici A, Kuru O. Reliability and validity of the Turkish version of the Falls Efficacy Scale International (FES-I) in community-dwelling older persons. Arch Gerontol Geriatr. 2012 May-Jun;54(3):429-33. doi: 10.1016/j.archger.2011.06.010. Epub 2011 Aug 9. PMID 21831462
- [Background] Delbaere K, Close JC, Mikolaizak AS, Sachdev PS, Brodaty H, Lord SR. The Falls Efficacy Scale International (FES-I). A comprehensive longitudinal validation study. Age Ageing. 2010 Mar;39(2):210-6. doi: 10.1093/ageing/afp225. Epub 2010 Jan 8. PMID 20061508
- [Background] Beaudart C, Biver E, Reginster JY, Rizzoli R, Rolland Y, Bautmans I, Petermans J, Gillain S, Buckinx F, Van Beveren J, Jacquemain M, Italiano P, Dardenne N, Bruyere O. Development of a self-administrated quality of life questionnaire for sarcopenia in elderly subjects: the SarQoL. Age Ageing. 2015 Nov;44(6):960-6. doi: 10.1093/ageing/afv133. Epub 2015 Oct 3. PMID 26433796
- [Background] Erdogan T, Eris S, Avci S, Oren MM, Kucukdagli P, Kilic C, Beaudart C, Bruyere O, Karan MA, Bahat G. Sarcopenia quality-of-life questionnaire (SarQoL)(R): translation, cross-cultural adaptation and validation in Turkish. Aging Clin Exp Res. 2021 Nov;33(11):2979-2988. doi: 10.1007/s40520-020-01780-0. Epub 2021 Feb 4. PMID 33538991
- [Background] Rodrigues A, Janssens L, Langer D, Matsumura U, Rozenberg D, Brochard L, Reid WD. Semi-automated Detection of the Timing of Respiratory Muscle Activity: Validation and First Application. Front Physiol. 2022 Jan 3;12:794598. doi: 10.3389/fphys.2021.794598. eCollection 2021. PMID 35046839
- [Background] Illi SK, Held U, Frank I, Spengler CM. Effect of respiratory muscle training on exercise performance in healthy individuals: a systematic review and meta-analysis. Sports Med. 2012 Aug 1;42(8):707-24. doi: 10.1007/BF03262290. PMID 22765281
- [Background] Zeren M, Cakir E, Gurses HN. Effects of inspiratory muscle training on postural stability, pulmonary function and functional capacity in children with cystic fibrosis: A randomised controlled trial. Respir Med. 2019 Mar;148:24-30. doi: 10.1016/j.rmed.2019.01.013. Epub 2019 Jan 28. PMID 30827470